CLINICAL TRIAL: NCT04114630
Title: A 12-month Prospective, Phase IIIb, Multicenter, Open-label Clinical Trial to Assess Health-related Quality of Life (HRQoL) in Patients With Chronic or High-frequency Episodic Migraine Treated With Erenumab Who Present Associated Comorbidities
Brief Title: Study of Quality of Life in Subjects With Chronic or High-frequency Episodic Migraine and Associated Comorbidities Treated With Erenumab
Acronym: COMIG
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: No patients were enrolled and global prioritization of pipeline and research strategy
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CAMG334AES01; 2019-001820-36 (EudraCT Number)
Record Dates: First submitted 2019-08-21; First posted 2019-10-03 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2019-09

CONDITIONS: Migraine
Keywords: Chronic migraine; Migraine; Transformative migraine; Neurologic disease; Unremitting pain; Progressive over time; Nausea; Vomiting; Sensitivity to light,; Sensitivity to sound; Pain localized to one side of head,; Painful headache; Pain in head; Head throbbing; Sinus headache; Pounding headache
MeSH Terms: conditions — Migraine Disorders; Nausea; Vomiting; Photophobia; Headache | interventions — erenumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- erenumab (Experimental): Solution for s.c injection. Prefilled autoinjector
  Interventions: Drug: erenumab 70mg/mL

INTERVENTIONS:
Drug: erenumab 70mg/mL — Unit dose: 70 mg/mL single-dose., prefilled erenumab autoinjectors. 140 mg dose = 2 x 70 mg/mL, single dose, prefilled erenumab autoinjectors
  Other Names: AMG334

SUMMARY:
Migraine is a very common, neurological disorder, characterized by recurrent episodes of headache, potential progression to more frequent and severe attack patterns, and associated symptoms. In Spain, the prevalence rates are 12-13% and in women up to 17-18% Migraine has been shown to largely impair patient's Health-Related Quality of Life (HRQoL), affecting work, household chores, social activities and family life. Recurrent headache attacks and frequently persistent fear and concern about the next attack disrupt the patient's familial, occupational and social life, and reduce his/her expectations for career and financial future. The consequences of this loss of productivity is also shared in his/her private life with their family. For this reason, not only the clinical benefit but other dimensions as HRQoL or work affectation should be added to the study of the benefits of migraine treatment.

Migraine pathophysiology pathways may be shared with other illness, such as fibromyalgia, chronic fatigue or Irritable Bowel Syndrome (IBS) . The purpose of the present clinical trial is to evaluate whether erenumab, at a target dose of 70 mg or 140 mg for a period of 12 months, impacts Health-Related Quality of Life (HRQoL) among patients withchronic migraine (CM) or High-Frequency Episodic Migraine (HFEM) who are affected with at least one comorbidity (fibromyalgia, fatigue and IBS). Data from this study, will provide additional information to help clinicians in treating patients with migraine and other illness.

ELIGIBILITY:
Inclusion Criteria: key inclusion citeria

During the Screening Epoch:

1. Signed informed consent must be obtained prior to participation in the study.
2. Adults ≥18 years of age upon entry into screening.
3. Patient diagnosed with chronic and high -frequency episodic migraine (with or without aura) for at least 1 year prior to screening according to the International Classification of Headache Disorders-3rd Edition (ICHD-3).
4. Patient with a documented diagnosis in clinical history of one or more of the following comorbidities: chronic fatigue, fibromyalgia and/or IBS.
5. Patients previously treated with other monoclonal antibodies for migraine can be included if the appropriate washout period according to product half-life has been done for each monoclonal antibody.

During the Baseline Epoch:

1. Migraine frequency of ≥ 10 migraine days during the Baseline Epoch, confirmed by the eDiary.
2. ≥ 80% eDiary compliance during the Baseline Epoch.

Exclusion Criteria: Key Exclusion criteria

1. Older than 50 years of age at migraine onset.
2. Unable to differentiate migraine from other headaches.
3. History of cluster headache or hemiplegic migraine headache.
4. Used a device, or procedure within 2 months prior to the start of or during baseline or during the treatment period.
5. Use of other investigational drugs within 5 half-lives of enrollment or inappropriate washout period in case of monoclonal antibodies, or until the expected pharmacodynamic effect has returned to baseline, whichever is longer.
6. Unlikely to be able to complete all protocol required study visits or procedures, and/or to comply with all required study procedures.
7. History or evidence of any other unstable or clinically significant medical condition that in the opinion of the investigator would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion.

Other protocol-defined inclusion/exclusion criteria may apply at the end.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-30 (Estimated); Primary Completion 2021-12-06 (Estimated); Study Completion 2022-01-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients (in the overall population and by each comorbidity) who achieve a ≥5-point increase in the MSQ-RFR, MSQ-RFP domains and a ≥8-point increase in the MSQ-EF domain of the Migraine-Specific Quality of Life Questionnaire (MSQ 2.1) | Baseline up to approximately 12 months
  MSQ 2.1 consists of 14 items that address 3 domains:(1) Role Function-Restrictive (items 1-7);(2) Role Function- Preventive (items 8-11);&(3) Emotional Function (items 12-14).Response options range from "none of the time" (value 1) to "all of the time" (value 6), & are reverse-recoded (value 6 to 1) before the domain scores are calculated.Total raw scores for each domain is the sum of the final item value for all of the items in that domain.After the total raw score is computed for each domain, they are transformed to a 0-100 scale with higher scores indicating a better health status & a positive change in scores reflecting functional improvement. Comorbidities include fibromyalgia, chronic fatigue, and/or irritable bowel syndrome (IBS)

SECONDARY OUTCOMES:
Association between MSQ 2.1 and other HRQoL scores in each comorbidity (fibromyalgia, chronic fatigue, and/or IBS). | Baseline, month 3, 6 and 12.
  Correlation between HRQoL scores in migraine questionnaire (MSQ 2.1) and HRQoL scores in each comorbidity questionnaire: fibromyalgia (Fibromyalgia Impact Questionnaire, FIQ), chronic fatigue (Short Form health survey, SF-12) and IBS (Irritable Bowel Syndrome Quality of Life, IBS-QOL) in all study visits.
Mean change in HRQoL | Baseline, month 6 and 12.
  Health Related Quality of Life (HRQoL) in patients with migraine and at least once of these comorbitiy (fibromyalgia, chronic fatigue and irritable bowel syndrome [IBS])
Patient profile: number of migraine episodes/month | Baseline
  This description can help to understand the baseline characteristics of patients treated with erenumab and the relation with the outcomes
Duration and exposure of 70 and 140 mg doses of erenumab | Baseline up to approximately 1 year
  Dosing information will be collected throughout the trial including dose modifications and missed doses to provide total exposure of drug over time.
Change in the mean number of migrane days per month from baseline to month 12 | From baseline to month 12
  • Efficacy of erenumab will be assessed by migraine days.
Change in the mean number of days of use of acute migraine-specific medication per month from baseline to month 12 | From baseline to month 12.
  • Efficacy of erenumab.
Percentage of patients who achieve at least 50% or greater reduction in the mean number of migraine days per month from baseline to month 12. | From baseline to month 12
  • Efficacy of erenumab.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (23):
- Spain (23):
  - Novartis Investigative Site, Seville, Andalicía
  - Novartis Investigative Site, Cadiz, Andalusia
  - Novartis Investigative Site, Córdoba, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Zaragoza, Aragon
  - Novartis Investigative Site, Palma de Mallorca, Balearic Islands
  - Novartis Investigative Site, Barakaldo, Basque Country
  - Novartis Investigative Site, Bilbao, Basque Country
  - Novartis Investigative Site, Santa Cruz de Tenerife, Canary Islands
  - Novartis Investigative Site, Valladolid, Castille and León
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, Lugo, Galicia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Alcorcón, Madrid
  - Novartis Investigative Site, Fuenlabrada, Madrid
  - Novartis Investigative Site, Pozuelo de Alarcón, Madrid
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, Elda, Valencia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigational Site, Valencia, Valencia
  - Novartis Investigative Site, Madrid
  - Novartis Investigatice Site, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com